CLINICAL TRIAL: NCT01812044
Title: Postoperative Subtenons Anesthesia for Postoperative Pain in Pediatric Strabismus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Pro00033000
Record Dates: First submitted 2013-03-13; First posted 2013-03-15 (Estimated); Results first posted 2016-04-26 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-03

CONDITIONS: Strabismus
MeSH Terms: conditions — Strabismus | interventions — Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- subtenons anesthetic and topical control (Other): Group 1 (subtenons anesthetic and topical control): 0.5 cc of local anesthetic (preservative-free bupivacaine 0.75%) administered via a cannula subtenons through each surgical wound with 0.5 cc of Hypromellose 0.3% gel applied topically to each surgical wound at end of surgery
  Interventions: Drug: subtenons anesthetic - preservative-free bupivacaine 0.75%; Drug: topical control - 0.5 cc of Hypromellose 0.3% gel
- topical anesthetic and subtenons control (Other): Group 2 (topical anesthetic and subtenons control): 0.5 cc of lidocaine 3.5% ophthalmic gel applied topically to each surgical wound and 0.5 cc of normal saline (NS) administered via a cannula subtenons through each surgical wound at end of surgery
  Interventions: Drug: topical anesthetic - 0.5 cc of lidocaine 3.5% ophthalmic gel; Drug: subtenons control - 0.5 cc of Normal Saline
- topical control and subtenons control (Other): Group 3 (topical control and subtenons control): 0.5 cc of topical Hypromellose 0.3% gel applied topically to each surgical wound and 0.5 cc of NS administered via a cannula subtenons through each surgical wound at end of surgery
  Interventions: Drug: topical control - 0.5 cc of Hypromellose 0.3% gel; Drug: subtenons control - 0.5 cc of Normal Saline

INTERVENTIONS:
Drug: subtenons anesthetic - preservative-free bupivacaine 0.75%
  Arms: subtenons anesthetic and topical control
Drug: topical anesthetic - 0.5 cc of lidocaine 3.5% ophthalmic gel
  Arms: topical anesthetic and subtenons control
Drug: topical control - 0.5 cc of Hypromellose 0.3% gel
  Arms: subtenons anesthetic and topical control; topical control and subtenons control
Drug: subtenons control - 0.5 cc of Normal Saline
  Arms: topical anesthetic and subtenons control; topical control and subtenons control

SUMMARY:
The purpose of this study is to determine if local anesthetic, either a subtenons injection (an injection just beneath the surface tissue of the eye) or a topical ophthalmic gel (applied directly on the surface of the eye) given at the end of strabismus surgery reduces postoperative pain. Some surgeons routinely use either the subtenon and/or topical anesthetic for pain at the end of strabismus surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 year to < 8 years
* Undergoing strabismus surgery under general anesthesia
* No previous surgery on muscle to be operated
* No known allergy to lidocaine or bupivacaine
* Investigator willing to inject subtenons NS or preservative-free bupivacaine 0.75% by cannula into all surgical wounds and willing to administer topical lidocaine 3.5% ophthalmic gel or Hypromellose 0.3% gel (GenTeal Severe Dry Eye Relief) to all surgical wounds at the end of strabismus surgery.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Enyedi, MD, Principal Investigator — Duke Eye Center
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 57 participants signed consent. 7 participants were withdrawn by PI prior to randomization.
Groups:
- Subtenons Anesthetic and Topical Control: Group 1 (subtenons anesthetic and topical control): 0.5 cc of local anesthetic (preservative-free bupivacaine 0.75%) administered via a cannula subtenons through each surgical wound with 0.5 cc of Hypromellose 0.3% gel applied topically to each surgical wound at end of surgery
  subtenons anesthetic - preservative-free bupivacaine 0.75%
  topical control - 0.5 cc of Hypromellose 0.3% gel
- Topical Anesthetic and Subtenons Control: Group 2 (topical anesthetic and subtenons control): 0.5 cc of lidocaine 3.5% ophthalmic gel applied topically to each surgical wound and 0.5 cc of normal saline (NS) administered via a cannula subtenons through each surgical wound at end of surgery
  topical anesthetic - 0.5 cc of lidocaine 3.5% ophthalmic gel
  subtenons control - 0.5 cc of Normal Saline
- Topical Control and Subtenons Control: Group 3 (topical control and subtenons control): 0.5 cc of topical Hypromellose 0.3% gel applied topically to each surgical wound and 0.5 cc of NS administered via a cannula subtenons through each surgical wound at end of surgery
  topical control - 0.5 cc of Hypromellose 0.3% gel
  subtenons control - 0.5 cc of Normal Saline
Period: Overall Study
Arm/Group | Subtenons Anesthetic and Topical Control | Topical Anesthetic and Subtenons Control | Topical Control and Subtenons Control
Started | 17 | 17 | 16
Completed | 17 | 17 | 16
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subtenons Anesthetic and Topical Control | Topical Anesthetic and Subtenons Control | Topical Control and Subtenons Control | Total
Number analyzed (Participants) | 17 | 17 | 16 | 50
Age, Continuous [Mean (Full Range); unit: months] | 53.6 [13 to 87] | 50.1 [19 to 91] | 60.9 [27 to 89] | 54.9 [13 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 7 | 21
  Male | 10 | 10 | 9 | 29

OUTCOME MEASURES:

1. Primary Outcome: Average Pain Score Over the First 30 Post-operative Minutes Using the CHEOPS Scale
Description: Pain will be assessed by a masked observer using the Children's Hospital Eastern Ontario Pain Scale (CHEOPS) scale. The CHEOPS (Children's Hospital of Eastern Ontario Pain Scale) is a behavioral scale for evaluating postoperative pain in young children. The scale is assessed using the sum of a score for cry (1-3), facial expression (0-2), verbalization (0-2), torso (1-2), touch (1-2) and legs (1-2). The minimum score is 4, the maximum score is 13, and higher scores indicate more pain.
  Pain is rated every 5 minutes for the first 30 minutes postoperatively. Each pain score collected in the first 30 minutes was averaged to calculate a per per participant average pain score over the first 30 minutes . Then each participant's per participant average pain score was combined to calculate the reported mean for "Average pain score over the first 30 post-operative minutes using the CHEOPS scale." for each group.
Time Frame: 0-30 minutes post-operative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subtenons Anesthetic and Topical Control | Topical Anesthetic and Subtenons Control | Topical Control and Subtenons Control
Number analyzed (Participants) | 17 | 17 | 16
units on a scale | 6.36 (0.97) | 6.57 (1.06) | 6.58 (0.51)

2. Secondary Outcome: Peak Pain Score
Description: This secondary outcome will include the peak pain score for duration of follow up period. Pain will be assessed by masked observers, using the CHEOPS scale. The CHEOPS (Children's Hospital of Eastern Ontario Pain Scale) is a behavioral scale for evaluating postoperative pain in young children. The scale is assessed using the sum of a score for cry (1-3), facial expression (0-2), verbalization (0-2), torso (1-2), touch (1-2) and legs (1-2). The minimum score is 4, the maximum score is 13, and higher scores indicate more pain.
  A pain score was assessed and recorded every 5 minutes by a masked observer (clinical research coordinator) for the first 30 minutes after extubation, then every 15 minutes for the next hour, then, if applicable, hourly until discharge.
Time Frame: 0-150 minutes post-operative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subtenons Anesthetic and Topical Control | Topical Anesthetic and Subtenons Control | Topical Control and Subtenons Control
Number analyzed (Participants) | 17 | 17 | 16
units on a scale | 8.65 (2.42) | 10.47 (2.27) | 9.69 (2.15)
Statistical Analysis 1: Comparison: Subtenons Anesthetic and Topical Control vs Topical Anesthetic and Subtenons Control; Test type: Superiority or Other; p = 0.035, Wilcoxon (Mann-Whitney); P-value based on Wilcoxon rank sum test of difference in medians between groups
Statistical Analysis 2: Comparison: Subtenons Anesthetic and Topical Control vs Topical Control and Subtenons Control; Test type: Superiority or Other; p = 0.189, Wilcoxon (Mann-Whitney); P-value based on Wilcoxon rank sum test of difference in medians between groups
Statistical Analysis 3: Comparison: Topical Anesthetic and Subtenons Control vs Topical Control and Subtenons Control; Test type: Superiority or Other; p = 0.298, Wilcoxon (Mann-Whitney); P-value based on Wilcoxon rank sum test of difference in medians between groups

3. Secondary Outcome: Total Narcotic Use During Post-operative Recovery
Description: This secondary outcome will include total narcotic use
Time Frame: Total time in post-operative recovery - up to 6 hours
Measure: Mean (Standard Deviation); unit: mcg/kg
Arm/Group | Subtenons Anesthetic and Topical Control | Topical Anesthetic and Subtenons Control | Topical Control and Subtenons Control
Number analyzed (Participants) | 17 | 17 | 16
mcg/kg | 1.65 (0.61) | 1.78 (0.66) | 1.60 (.077)

4. Secondary Outcome: Negative Postoperative Behavior Score on the PHBQ (Post Hospitalization Behavioral Questionnaire)
Description: This secondary outcome will determine the negative postoperative behaviors based on the PHBQ questionnaire given to the parents of the child 1 week (+/- 3 days) post-operatively.
  with a score of 81 indicating no change, a score of less than 81 indicating a change for the better, and a score of over 81 indicating a change for the worse, on average, in behavior.
  Lowest score 27; highest score 135
Time Frame: 1 week (+/- 3 days) post operatively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subtenons Anesthetic and Topical Control | Topical Anesthetic and Subtenons Control | Topical Control and Subtenons Control
Number analyzed (Participants) | 17 | 17 | 16
units on a scale | 80.2 (7.8) | 78.2 (10.9) | 78.5 (12.1)

5. Secondary Outcome: Average Time to Discharge
Time Frame: 0-150 minutes post-operative
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Subtenons Anesthetic and Topical Control | Topical Anesthetic and Subtenons Control | Topical Control and Subtenons Control
Number analyzed (Participants) | 17 | 17 | 16
minutes | 106 (16) | 107 (25) | 106 (21)

6. Secondary Outcome: Number of Participants With Post Operative Nausea and Vomiting
Time Frame: 0-150 minutes post-operative
Measure: Number; unit: participants
Arm/Group | Subtenons Anesthetic and Topical Control | Topical Anesthetic and Subtenons Control | Topical Control and Subtenons Control
Number analyzed (Participants) | 17 | 17 | 16
participants | 1 | 1 | 1

7. Secondary Outcome: Number of Participants Who Required Anti-emetic Medication Post-operatively
Time Frame: Total time in post-operative recovery - up to 6 hours
Measure: Number; unit: participants
Arm/Group | Subtenons Anesthetic and Topical Control | Topical Anesthetic and Subtenons Control | Topical Control and Subtenons Control
Number analyzed (Participants) | 17 | 17 | 16
participants | 1 | 1 | 1

8. Secondary Outcome: Peak Pain Score During First 30 Minutes
Description: This secondary outcome will include the peak pain score for duration of follow up period. Pain will be assessed by masked observers, using the CHEOPS scale. The CHEOPS (Children's Hospital of Eastern Ontario Pain Scale) is a behavioral scale for evaluating postoperative pain in young children. The scale is assessed using the sum of a score for cry (1-3), facial expression (0-2), verbalization (0-2), torso (1-2), touch (1-2) and legs (1-2). The minimum score is 4, the maximum score is 13, and higher scores indicate more pain.
  Pain is rated every 5 minutes for the first 30 minutes postoperatively.
Time Frame: 0-30 minutes post-operative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subtenons Anesthetic and Topical Control | Topical Anesthetic and Subtenons Control | Topical Control and Subtenons Control
Number analyzed (Participants) | 17 | 17 | 16
units on a scale | 7.0 (1.9) | 7.8 (2.4) | 8.3 (2.7)

ADVERSE EVENTS:
Arm/Group | Subtenons Anesthetic and Topical Control | Topical Anesthetic and Subtenons Control | Topical Control and Subtenons Control
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes